CLINICAL TRIAL: NCT01482624
Title: Intra-articular Hyaluronan After Arthroscopic Meniscal Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VSK-BE-2011-11
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Arthroscopic Meniscal Surgery
Keywords: hyaluronan; hyaluronic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VISCOSEAL® SYRINGE (Active Comparator)
  Interventions: Device: Hyaluronan (0.5%, 5 mg/10 ml)
- Standard arthroscopic meniscal surgery (Other)
  Interventions: Procedure: Standard arthroscopic meniscal surgery

INTERVENTIONS:
Device: Hyaluronan (0.5%, 5 mg/10 ml) — Standard arthroscopic meniscal surgery and add-on treatment with VISCOSEAL® SYRINGE. Single injection of Hyaluronan directly after arthroscopic procedure.
  Arms: VISCOSEAL® SYRINGE
Procedure: Standard arthroscopic meniscal surgery — Standard arthroscopic meniscal surgery without add-on treatment.
  Arms: Standard arthroscopic meniscal surgery

SUMMARY:
The primary objective of this clinical investigation is to determine whether post-arthroscopic treatment with 10 ml of 0.5% sodium hyaluronate (VISCOSEAL® SYRINGE) can relief pain, improve mobility and promote joint recovery, compared to the standard arthroscopy procedure alone, in patients undergoing arthroscopic procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 75 years of age.
* Good general health condition.
* Signed written informed consent.
* Patients with necessity for arthroscopic meniscal surgery.
* Ensured compliance of subject over the whole study period.

Exclusion Criteria:

* Concomitant or previous participation in a clinical investigation within the last 3 months prior to study inclusion.
* Knee joint arthroscopy in study relevant joint within 6 months prior to study inclusion.
* Patients with known hypersensitivity to the investigational device (i.e. active compound and excipients) or any component or procedure used in the study.
* Contraindication for the use of the investigational product or for the scheduled arthroscopy, used anesthesia and post-surgical treatment.
* Concomitant disease of sufficient severity (e.g. uncontrolled diabetes mellitus, carcinoma, etc.), which in the opinion of the investigator, may put the patient at risk when participating in the study, or affect the patient's ability to take part in the study.
* Concomitant disease of sufficient severity at study relevant joint (e.g. known or suspected infection, peripheral neuropathy or presence of hemarthros).
* List of concomitant medications not allowed which interfere with the functional assessments of this study.
* Use of medication contraindicated for arthroscopic surgery.
* Intra-articular treatment with a sodium hyaluronate-based product within the last 6 months or use of corticosteroid containing substance within the last 3 months at study relevant joint.
* Recent history of drug and/or alcohol abuse (within the last 6 months) or patients with severe mental illness or suicidal tendency.
* Pregnant or lactating females.
* Participants of childbearing age (pre-menopausal) who do not accept the use of methods of birth control with pearl index ≤ 1% (i.e. oral contraceptives, vaginal ring, hormone-releasing Intrauterine Device (IUD), implants, depot syringes, hormone patch, double barrier method, tubal ligation, vasectomised partner,…) during the treatment period and the first 4 weeks of follow-up period.
* Subjects having a high probability of non-compliance to the study procedures according to investigator's judgement (like illiteracy, insufficient knowledge of local language).
* Kellgren III-IV on study relevant side (confirmed by X-ray).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pain evaluation (ordinal 11-point Likert scale) on day 84. | Day 84
  Intensity of pain will be evaluated on 11-point Likert ordinal scale ranging from '0' (no pain) to '10' (extreme pain).

SECONDARY OUTCOMES:
Pain evaluation (ordinal 11-point Likert scale) on day of arthroscopy. | Day 0
  Intensity of pain will be evaluated on 11-point Likert ordinal scale ranging from '0' (no pain) to '10' (extreme pain).
Pain evaluation (ordinal 11-point Likert scale) on day 14. | Day 14
  Intensity of pain will be evaluated on 11-point Likert ordinal scale ranging from '0' (no pain) to '10' (extreme pain).
Pain evaluation (ordinal 11-point Likert scale) on day 42. | Day 42
  Intensity of pain will be evaluated on 11-point Likert ordinal scale ranging from '0' (no pain) to '10' (extreme pain).
Patient's and investigator's global evaluation of study-relevant knee complaints on day 14. | On Day 14
  Measured by Clinical Global Impression (CGI) 7-point scale, ranking from 'very much improved' to 'very much worse' condition.
Patient's and investigator's global evaluation of study-relevant knee complaints on day 42. | On Day 42
  Measured by Clinical Global Impression (CGI) 7-point scale, ranking from 'very much improved' to 'very much worse' condition.
Patient's and investigator's global evaluation of study-relevant knee complaints on day 84. | On Day 84
  Measured by Clinical Global Impression (CGI) 7-point scale, ranking from 'very much improved' to 'very much worse' condition.
Range of Motion at baseline. | Baseline
  Range of Motion of the study relevant knee will be evaluated by a handheld goniometer using the Neutral-0-Method. Measurement unit: degree.
Range of Motion on day of arthroscopy. | On Day 0
  Range of Motion of the study relevant knee will be evaluated by a handheld goniometer using the Neutral-0-Method. Measurement unit: degree.
Range of Motion on day 14. | On Day 14
  Range of Motion of the study relevant knee will be evaluated by a handheld goniometer using the Neutral-0-Method. Measurement unit: degree.
Range of Motion on day 42. | On Day 42
  Range of Motion of the study relevant knee will be evaluated by a handheld goniometer using the Neutral-0-Method. Measurement unit: degree.
Range of Motion on day 84. | On Day 84
  Range of Motion of the study relevant knee will be evaluated by a handheld goniometer using the Neutral-0-Method. Measurement unit: degree.
Walking ability on day of arthroscopy. | On Day 0
  Patient's walking ability will be evaluated with respect to difficulty on walking 100 metres and pain on walking 100 metres.
  Measured by 5-point scale, ranking from 'none' to 'extreme' difficulty.
Walking ability on day 14. | On Day 14
  Patient's walking ability will be evaluated with respect to difficulty on walking 100 metres and pain on walking 100 metres.
  Measured by 5-point scale, ranking from 'none' to 'extreme' difficulty.
Walking ability on day 42. | On Day 42
  Patient's walking ability will be evaluated with respect to difficulty on walking 100 metres and pain on walking 100 metres.
  Measured by 5-point scale, ranking from 'none' to 'extreme' difficulty.
Walking ability on day 84. | On Day 84
  Patient's walking ability will be evaluated with respect to difficulty on walking 100 metres and pain on walking 100 metres.
  Measured by 5-point scale, ranking from 'none' to 'extreme' difficulty.
Health-related quality of life questionnaire at baseline. | At baseline
  The descriptive system of health-related quality of life states consists of five dimensions:
  * Mobility,
  * Self-Care,
  * Usual Activities,
  * Pain/Discomfort,
  * Anxiety/Depression.
  The responses record three levels of severity (no problems/some or moderate problems/extreme problems).
  For recording the individual's rating for their current health-related quality of life state, a standard vertical 20 cm visual analogue scale (similar to a thermometer) is utilised.
Health-related quality of life questionnaire on day of arthroscopy. | On day 0
  The descriptive system of health-related quality of life states consists of five dimensions:
  * Mobility,
  * Self-Care,
  * Usual Activities,
  * Pain/Discomfort,
  * Anxiety/Depression.
  The responses record three levels of severity (no problems/some or moderate problems/extreme problems).
  For recording the individual's rating for their current health-related quality of life state, a standard vertical 20 cm visual analogue scale (similar to a thermometer) is utilised.
Health-related quality of life questionnaire on day 14. | On day 14
  The descriptive system of health-related quality of life states consists of five dimensions:
  * Mobility,
  * Self-Care,
  * Usual Activities,
  * Pain/Discomfort,
  * Anxiety/Depression.
  The responses record three levels of severity (no problems/some or moderate problems/extreme problems).
  For recording the individual's rating for their current health-related quality of life state, a standard vertical 20 cm visual analogue scale (similar to a thermometer) is utilised.
Health-related quality of life questionnaire on day 42. | On day 42
  The descriptive system of health-related quality of life states consists of five dimensions:
  * Mobility,
  * Self-Care,
  * Usual Activities,
  * Pain/Discomfort,
  * Anxiety/Depression.
  The responses record three levels of severity (no problems/some or moderate problems/extreme problems).
  For recording the individual's rating for their current health-related quality of life state, a standard vertical 20 cm visual analogue scale (similar to a thermometer) is utilised.
Health-related quality of life questionnaire on day 84. | On day 84
  The descriptive system of health-related quality of life states consists of five dimensions:
  * Mobility,
  * Self-Care,
  * Usual Activities,
  * Pain/Discomfort,
  * Anxiety/Depression.
  The responses record three levels of severity (no problems/some or moderate problems/extreme problems).
  For recording the individual's rating for their current health-related quality of life state, a standard vertical 20 cm visual analogue scale (similar to a thermometer) is utilised.
Joint Examination Parameters at baseline. | At baseline
  Joint Examination comprises
  * Intensity of effusion (measured by 5-point scale, ranking from 'none' to 'extreme' intensity),
  * Necessity of puncture,
  * Clinical parameters: redness, warmth, swelling, tenderness on palpation (measured by 5-point Likert scale, ranging from 'none' to 'extreme' intensity).
Joint Examination Parameters on day of arthroscopy. | On Day 0
  Joint Examination comprises
  * Intensity of effusion (measured by 5-point scale, ranking from 'none' to 'extreme' intensity),
  * Necessity of puncture,
  * Clinical parameters: redness, warmth, swelling, tenderness on palpation (measured by 5-point Likert scale, ranging from 'none' to 'extreme' intensity).
Joint Examination Parameters on day 14. | On Day 14
  Joint Examination comprises
  * Intensity of effusion (measured by 5-point scale, ranking from 'none' to 'extreme' intensity),
  * Necessity of puncture,
  * Clinical parameters: redness, warmth, swelling, tenderness on palpation (measured by 5-point Likert scale, ranging from 'none' to 'extreme' intensity).
Joint Examination Parameters on day 42. | On Day 42
  Joint Examination comprises
  * Intensity of effusion (measured by 5-point scale, ranking from 'none' to 'extreme' intensity),
  * Necessity of puncture,
  * Clinical parameters: redness, warmth, swelling, tenderness on palpation (measured by 5-point Likert scale, ranging from 'none' to 'extreme' intensity).
Joint Examination Parameters on day 84. | On Day 84
  Joint Examination comprises
  * Intensity of effusion (measured by 5-point scale, ranking from 'none' to 'extreme' intensity),
  * Necessity of puncture,
  * Clinical parameters: redness, warmth, swelling, tenderness on palpation (measured by 5-point Likert scale, ranging from 'none' to 'extreme' intensity).
Frequency of test product-related Adverse Events | Up to Day 84
Pain evaluation (ordinal 11-point Likert scale) at baseline. | Baseline
  Intensity of pain will be evaluated on 11-point Likert ordinal scale ranging from '0' (no pain) to '10' (extreme pain).
Walking ability at baseline. | Baseline
  Patient's walking ability will be evaluated with respect to difficulty on walking 100 metres and pain on walking 100 metres.
  Measured by 5-point scale, ranking from 'none' to 'extreme' difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Roger van Riet, MD, Principal Investigator — AZ Monica, Orthopedisch centrum SPM, Deurne (Belgium)
Locations (1):
- AZ Monica, Orthopedisch centrum SPM, Deurne, Belgium